CLINICAL TRIAL: NCT04423510
Title: Previously Operated Recurrent Pilonidal Sinus Treated With Crystallized Phenol: Twenty Years Experience
Brief Title: Nonoperative Treatment of Recurrent Pilonidal Sinus Disease
Status: Completed | Type: Observational
Sponsor: Osman DOĞRU (Other)
Responsible Party: Sponsor-Investigator, Osman DOĞRU, Professor, MD, Konya Meram State Hospital
Organization: Konya Meram State Hospital (Other)
Other Study IDs: KonyaTRH01
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Pilonidal Sinus
Keywords: recurrent pilonidal disease; nonoperative treatment; crystallized phenol
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Recurrent pilonidal sinus: Postoperative recurrent pilonidal sinus disease
  Interventions: Procedure: Crystallized phenol treatment

INTERVENTIONS:
Procedure: Crystallized phenol treatment

SUMMARY:
Postoperative recurrent pilonidal sinus disease is troublesome and its treatment is challenge. Many treatment modalities have been advocated in the treatment of recurrent pilonidal sinus disease; however, there is still no consensus in the literature. Some minimally invasive techniques are used alone or as an adjunct to surgery. Crystallized phenol is the most popular method in the nonoperative treatment of primer pilonidal sinus disease. But its long term effect in the postoperative recurrent cases is unclear. Investigators aimed to present the long-term efficacy of crystallized phenol treatment on postoperative recurrent pilonidal sinus disease through our results collected within the last 20 years.

DETAILED DESCRIPTION:
Study data were collected prospectively and analyzed retrospectively. The demographic data of the patients, other parameters such as smoking, whether they sit a lot due to occupation (sitting at work for at least 6 hours a day), skin tone (whiter, darker), presence of positive family history, BMI (kg/m2, patients were divided into BMI <30 and BMI> 30), pilosity levels (mild,moderate, severe) were also recorded. In addition, the time from the recurrence to admission, the number and type of previous operations, and the status of the sinus at presentation (acute, chronic) were recorded. The presence of purulent discharge from the sinus opening and the presence of signs of inflammation or abscess formation in this region were evaluated as acute pilonidal sinus disease (PSD). The presence of serous discharge from the sinus opening and absence of abscess formation were evaluated as chronic PSD. Investigators investigated whether the factors mentioned above affect the number of applications and recurrence after crystallized phenol treatment (CPT).

The treatment procedure was applied to all patients by one surgical team. One day before the procedure, patients were asked to clean the hair from the waist to the middle of the thighs with depilatory creams or epilation. After local anesthesia was performed around the holes, a thin mosquito clamp was inserted into the sinus and the hairs were removed and the skin around the hole was covered by nitrofurantoin pomade to prevent chemical irritation. Then crystallized phenol was introduced into the sinus with the same clamp. Patients were allowed to return to their daily activities after the procedure. This procedure was performed every 3 weeks. If there was discharge from the wound during the follow-up examination, the procedure was repeated. The closure of the sinus hole and the complete disappearance of the discharge were accepted as healing. After the treatment, follow-up was started. Follow up was done first yearly than five years intervals. All of our patients' contact information was recorded by us and we tried to reach the patients every 5 years by any means (phone or e-mail). Investigators tried to follow them up by contacting them periodically, whether they contact us or not. According to this follow-up, patients were analyzed by divided into 3 groups(1-5 years, 5-10 years, 10-20 years). Patients who could not be reached by any means of communication were included in the unreachable group. Patients were recommended to have hair removal at the wound site once a month for 6 years.

Number of crystallized phenol application, presence of recurrence and number of recurrence after CPT and follow-up data were evaluated. Recurrence of the sinus hole which was found to occur again at least 6 months after being determined to be closed was considered as recurrence. If no recurrence was observed during the follow-up or if post-CPT recurrence was healed after treatment, CPT was considered successful.

ELIGIBILITY:
Inclusion Criteria:

* Previous operated recurrent pilonidal sinus disease
* Follow-up period of more than 12 months
* The patients who connection by e-mail or telephone

Exclusion Criteria:

* Primer pilonidal sinus disease
* Follow-up period of less than 12 months
* The patients who can't connection by e-mail or telephone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who previous operated recurrent pilonidal sinus disease and who accepted crystallized phenol treatment were included in the study. Patients who at least one year of treatment and contacting later were included in our study.
Sampling Method: Probability Sample
Enrollment: 227 (Actual)
Dates: Start 1995-03-01 (Actual); Primary Completion 2015-02-01 (Actual); Study Completion 2016-02-01 (Actual)

PRIMARY OUTCOMES:
Long term effect of crystallized phenol treatment in recurrent pilonidal sinus | January 1995-February 2015
  All participants we applied to crystallized phenol treatment (CPT) were contacted via e-mail, telephone or face-to-face interview and questioned whether there was a recurrence. The number of CPT applications and sinus characteristics (primer openings, seconder openings, sinus presentation etc.) were compared between recurrent participants and non-recurrent participants. The number of CPT application and sinus characteristic features was obtained patients files that were recorded in first consult.

SECONDARY OUTCOMES:
The effects of factors playing a role in the etiology of pilonidal sinus on treatment results | January 1995-February 2016
  All participants we applied to crystallized phenol treatment were contacted via e-mail, telephone or face-to-face interview and questioned whether there was a recurrence. The relationship between relapsed participants and non-relapsed participants was investigated between the factors accused in etiology (gender, BMI, family history, pilosity levels, skin tone etc.). Factors accused in etiology were obtained patients files that were recorded in first consult.

CONTACTS AND LOCATIONS:
Overall Officials: Ersin TURAN, 3, Study Chair — Konya Education and Research Hospital; Ramazan Saygın KERİMOĞLU, 4, Study Chair — Konya Education and Research Hospital; Emet Ebru NAZİK, 5, Study Chair — Konya Education and Research Hospital; Ebru Esen, 6, Study Chair — Konya Education and Research Hospital

IPD SHARING:
Plan to Share IPD: Yes
We are planned to share that all of individual participant data.
Supporting Information: SAP, ICF
Time Frame: The data will become available starting 6 months after publication.
Access Criteria: The data will share as SPSS dataset.

REFERENCES:
- [Background] Lund JN, Leveson SH. Fibrin glue in the treatment of pilonidal sinus: results of a pilot study. Dis Colon Rectum. 2005 May;48(5):1094-6. doi: 10.1007/s10350-004-0905-4. PMID 15868239
- [Background] Dessily M, Charara F, Ralea S, Alle JL. Pilonidal sinus destruction with a radial laser probe: technique and first Belgian experience. Acta Chir Belg. 2017 Jun;117(3):164-168. doi: 10.1080/00015458.2016.1272285. Epub 2017 Jan 6. PMID 28056720
- [Background] Othman I. Skin glue improves outcome after excision and primary closure of sacrococcygeal pilonidal disease. Indian J Surg. 2010 Dec;72(6):470-4. doi: 10.1007/s12262-010-0170-9. Epub 2010 Nov 16. PMID 22131657
- [Result] Stauffer VK, Luedi MM, Kauf P, Schmid M, Diekmann M, Wieferich K, Schnuriger B, Doll D. Common surgical procedures in pilonidal sinus disease: A meta-analysis, merged data analysis, and comprehensive study on recurrence. Sci Rep. 2018 Feb 15;8(1):3058. doi: 10.1038/s41598-018-20143-4. PMID 29449548
- [Result] Doll D, Luedi MM, Wysocki AP. Pilonidal sinus disease guidelines: a minefield? Tech Coloproctol. 2016 Apr;20(4):263-4. doi: 10.1007/s10151-015-1398-y. Epub 2015 Dec 17. No abstract available. PMID 26681445
- [Result] Dag A, Colak T, Turkmenoglu O, Sozutek A, Gundogdu R. Phenol procedure for pilonidal sinus disease and risk factors for treatment failure. Surgery. 2012 Jan;151(1):113-7. doi: 10.1016/j.surg.2011.07.015. Epub 2011 Oct 6. PMID 21982072
- [Result] Kaymakcioglu N, Yagci G, Simsek A, Unlu A, Tekin OF, Cetiner S, Tufan T. Treatment of pilonidal sinus by phenol application and factors affecting the recurrence. Tech Coloproctol. 2005 Apr;9(1):21-4. doi: 10.1007/s10151-005-0187-4. PMID 15868494
- [Result] Dogru O, Camci C, Aygen E, Girgin M, Topuz O. Pilonidal sinus treated with crystallized phenol: an eight-year experience. Dis Colon Rectum. 2004 Nov;47(11):1934-8. doi: 10.1007/s10350-004-0720-y. PMID 15622588
- [Result] Aygen E, Arslan K, Dogru O, Basbug M, Camci C. Crystallized phenol in nonoperative treatment of previously operated, recurrent pilonidal disease. Dis Colon Rectum. 2010 Jun;53(6):932-5. doi: 10.1007/DCR.0b013e3181d8283b. PMID 20485008
- [Result] Emiroglu M, Karaali C, Esin H, Akpinar G, Aydin C. Treatment of pilonidal disease by phenol application. Turk J Surg. 2017 Mar 1;33(1):5-9. doi: 10.5152/UCD.2016.3532. eCollection 2017. PMID 28589180